CLINICAL TRIAL: NCT00005090
Title: A Randomized Phase III Trial Comparing Early High Dose Chemotherapy and an Autologous Stem Cell Transplant to Conventional Dose ABVD Chemotherapy for Patients With Advanced Stage Poor Prognosis Hodgkin's Disease as Defined by the International Prognostic Factors Project on Advanced Hodgkin's Disease
Brief Title: S9901 Combination Chemotherapy With or Without Peripheral Stem Cell Transplantation in Treating Men With Stage III or Stage IV Hodgkin's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: poor accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067708; S9901 (Other: SWOG); CLB-59802 (Other: CALGB); E-S9901 (Other: ECOG); U10CA032102 (NIH)
Record Dates: First submitted 2000-04-06; First posted 2003-08-28 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Lymphoma
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bleomycin; Carmustine; Cyclophosphamide; Dacarbazine; Doxorubicin; Etoposide; Vinblastine; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABVD x 5 + ABVD x 3 (Active Comparator): Patients receive 5 28-day cycles of ABVD (doxorubicin 25 mg/m^2, bleomycin 10 U/m^2, vinblastine 6 mg/m^2, dacarbazine 375 mg/m^2 all on days 1 and 15). Patients with no disease progression are then randomized to either 3 more cycles of ABVD or 1 more cycle of ABVD + high-dose therapy + stem cell transplant.
  Interventions: Biological: bleomycin sulfate; Drug: dacarbazine; Drug: doxorubicin hydrochloride; Drug: vinblastine
- ABVD x 5 + ABVD x 1 + HDT + PBSCT (Experimental): Patients receive 5 28-day cycles of ABVD (doxorubicin 25 mg/m^2, bleomycin 10 U/m^2, vinblastine 6 mg/m^2, dacarbazine 375 mg/m^2 all on days 1 and 15). Patients with no disease progression are then randomized to either 3 more cycles of ABVD or 1 more cycle of ABVD + high-dose therapy + stem cell transplant. Patients randomized to the transplant arm have 2 x 10^6 CD34+ blood mononuclear cells/kg of actual body weight collected at day -7. High dose therapy consists of BCNU 150/m^2 on days -6 to -4, etoposide 60 mg/kg on day -4, and cyclophosphamide 100 mg/kg on day -2. Peripheral blood stem cells are infused on day 0.
  Interventions: Biological: bleomycin sulfate; Drug: carmustine; Drug: cyclophosphamide; Drug: dacarbazine; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: vinblastine; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: bleomycin sulfate — 10 U/m^2 given on days 1 and 15 for 5 28-day cycles of ABVD. Patients with no disease progression are then randomized to either 3 more cycles of ABVD or 1 more cycle of ABVD + high-dose therapy + stem cell transplant.
Drug: carmustine — 150/m^2 on days -6 to -4 (4-6 days before transplant).
  Other Names: BCNU
  Arms: ABVD x 5 + ABVD x 1 + HDT + PBSCT
Drug: cyclophosphamide — 100 mg/kg on day -2 (2 days before transplant).
  Arms: ABVD x 5 + ABVD x 1 + HDT + PBSCT
Drug: dacarbazine — 375 mg/m^2 on days 1 and 15 for 5 28-day cycles of ABVD. Patients with no disease progression are then randomized to either 3 more cycles of ABVD or 1 more cycle of ABVD + high-dose therapy + stem cell transplant.
Drug: doxorubicin hydrochloride — 25 mg/m^2 on days 1 and 15 for 5 28-day cycles of ABVD. Patients with no disease progression are then randomized to either 3 more cycles of ABVD or 1 more cycle of ABVD + high-dose therapy + stem cell transplant.
Drug: etoposide — 60 mg/kg on day -4 (4 days before transplant).
  Arms: ABVD x 5 + ABVD x 1 + HDT + PBSCT
Drug: vinblastine — 6 mg/m^2 on days 1 and 15 for 5 28-day cycles of ABVD. Patients with no disease progression are then randomized to either 3 more cycles of ABVD or 1 more cycle of ABVD + high-dose therapy + stem cell transplant.
Procedure: peripheral blood stem cell transplantation — 2 x 10^6 CD34+ blood mononuclear cells/kg of actual body weight
  Arms: ABVD x 5 + ABVD x 1 + HDT + PBSCT

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. It is not yet known if combination chemotherapy is more effective with or without peripheral stem cell transplantation in treating Hodgkin's Disease.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without peripheral stem cell transplantation in treating men who have stage III or stage IV Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare progression-free and overall survival of patients with stage III or IV Hodgkin's disease treated with doxorubicin, bleomycin, vinblastine, and dacarbazine with or without autologous peripheral blood stem cell transplantation and high-dose chemotherapy.
* Compare the toxic effects of these treatment regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to number of poor prognostic factors (3 vs 4 vs 5) and stage of disease (III vs IV).

Patients receive induction chemotherapy consisting of doxorubicin IV over 5 minutes, bleomycin IV over 10 minutes, vinblastine IV over 5 minutes, and dacarbazine IV over 15-30 minutes on days 1 and 15. Treatment repeats every 28 days for 5 courses in the absence of disease progression or unacceptable toxicity. Patients who show at least partial response after the fifth course of induction chemotherapy and whose blood counts have recovered are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive 3 additional courses of induction chemotherapy for a total of 8 courses.
* Arm II: Patients receive 1 additional course of induction chemotherapy followed by stem cell collection. Patients then receive high-dose chemotherapy with carmustine IV over 2 hours on days -6 to -4, etoposide IV over 4 hours on day -4, and cyclophosphamide IV on day -2. Patients undergo autologous peripheral blood stem cell transplantation on day 0.

Patients are followed at 60 days, every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 460 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage III or IV Hodgkin's disease with at least 3 of the following characteristics:

  * Albumin less than 4.0 mg/dL
  * Hemoglobin less than 10.5 g/dL
  * Leukocytosis at least 15,000/mm^3
  * Lymphocytopenia less than 600/mm^3 or less than 8% of total WBC
  * Male sex
  * At least 45 years of age
  * Stage IV disease
* Bidimensionally measurable disease
* Bilateral or unilateral bone marrow aspiration and biopsy performed within 42 days of study
* Negative chest x-ray within 42 days of study OR
* Chest x-ray performed within 28 days of study
* Negative CT scan of thorax, abdomen, and pelvis within 42 days of study OR
* CT scan of thorax, abdomen, and pelvis performed within 28 days of study
* No history of lymphoma, myelodyplastic syndrome, or leukemia
* No CNS involvement by Hodgkin's disease

PATIENT CHARACTERISTICS:

Age:

* 15 to 65

Performance status:

* Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* See Disease Characteristics
* Bilirubin no greater than 1.5 times upper limit of normal (ULN) (unless elevation due to liver infiltration by Hodgkin's disease)
* Lymphoma-related hepatic dysfunction allowed

Renal:

* Creatinine no greater than 2.0 times ULN
* Creatinine clearance at least 60 mL/min
* Lymphoma-related renal dysfunction allowed

Cardiovascular:

* No coronary artery disease, cardiomyopathy, congestive heart failure, or arrhythmias requiring therapy
* Ejection fraction normal
* No significant EKG abnormalities suggesting active cardiac disease

Pulmonary:

* Corrected DLCO at least 60% OR
* FEV1 at least 60% predicted

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No HIV or AIDS
* No other prior malignancy within past 5 years except adequately treated basal cell or squamous cell skin cancer
* No active bacterial, fungal, or viral infection*
* Afebrile for 3 consecutive days* NOTE: *Prior to randomization portion of study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for Hodgkin's disease except single course of ABVD (doxorubicin, bleomycin, vinblastine, and dacarbazine) within 35 days of study

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for Hodgkin's disease

Surgery:

* Not specified

Other:

* At least 3 days since prior antibiotics, antifungals, or antivirals (except for prophylactic therapy or fever associated with underlying lymphoma) (for randomization portion of study)

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2000-04; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | every 3 months while on protocol treatment, then every 6 months for 2 years, then annually thereafter

SECONDARY OUTCOMES:
overall survival | every 3 months while on treatment, then every 6 months thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R. Gaynor, MD, Study Chair — Loyola University; Sandra J. Horning, MD, Study Chair — Stanford University; Linda J. Burns, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (47):
- United States (47):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Schneider Children's Hospital at North Shore, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia